CLINICAL TRIAL: NCT04804007
Title: Randomized Phase 2 Trial of Maintenance Oral Etoposide or Observation Following High-dose Chemotherapy for Relapsed Metastatic Germ-Cell Tumor
Brief Title: Maintenance Oral Etoposide or Observation Following High-dose Chemo for GCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nabil Adra (Other)
Responsible Party: Sponsor-Investigator, Nabil Adra, Assistant Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0742
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Germ Cell Tumor; Non-seminomatous Germ Cell Tumor; Ovarian Germ Cell Tumor
Keywords: Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Nonseminomatous germ cell tumor | interventions — Etoposide

STUDY DESIGN:
Intervention Model Description: Patients who completed HDCT+PBSCT within the past 16 weeks will enroll and randomize in 1:1 fashion in blocks of 8 to maintenance daily oral etoposide 50mg vs. observation only.
  Randomization will be stratified based on:
  -Presence of platinum refractory disease status defined by radiographic or serologic progression within 4 weeks of first-line cisplatin-based combination chemotherapy: yes vs. no
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance Oral Etoposide (Experimental): Maintenance daily oral Etoposide.
  Interventions: Drug: Etoposide
- Observation (No Intervention): If randomized to Observation, subjects will jump to follow-up.

INTERVENTIONS:
Drug: Etoposide — etoposide will be provided with prescription for etoposide 50mg orally daily for 21 days out of 28 day cycles. Cycles will be repeated every 4 weeks for a total of 3 cycles.
  Arms: Maintenance Oral Etoposide

SUMMARY:
This is an open label randomized phase II trial of maintenance oral etoposide vs. observation in patinets with relapsed GCT treated with high-dose chemotherapy (HDCT) and peripheral-blood stem-cell transplant (PBSCT).

DETAILED DESCRIPTION:
This is a randomized phase 2 trial of maintenance etoposide versus observation following HDCT+PBSCT for relapsed GCT. Patients who completed HDCT+PBSCT within the past 16 weeks will enroll and randomize in 1:1 fashion to maintenance daily oral etoposide 50mg vs. observation only.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information
2. Age ≥ 18 years at the time of consent
3. Histological or serological evidence of non-seminomatous GCT
4. Relapsed disease after first-line cisplatin-based combination chemotherapy
5. Completed salvage treatment with HDCT and PBSCT for 2 tandem cycles per Institutional Guidelines
6. HDCT must have been used as the initial salvage chemotherapy regimen (2nd line therapy) 6.1. Note: 1 or 2 cycles of standard course regimens prior to HDCT are acceptable (regimens include VeIP [vinblastine+ifosfmaide+cisplatin] or TIP [paclitaxel+ifosfamide+cisplatin] or PVB [cisplatin+vinblastine+bleomycin]
7. Normal or declining tumor markers (AFP and hCG) at time of screening
8. Adverse events from prior therapy recovered to CTCAE v5.0 grade ≤ 2 at time of registration
9. Women with ovarian germ cell tumors are eligible
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 within 28 days of study registration
11. Last dose of HDCT must be ≤16 weeks from study registration
12. Adequate organ function lab values obtained within 28 days prior to study registration System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,000 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥8 g/dL Renal Serum creatinine <2mg/dL Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN

    AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR
    * 5 X ULN for subjects with liver metastases Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
13. If a female of childbearing potential, a negative urine pregnancy test within 28 days prior to receiving the first dose of study drug.

    o Non-childbearing potential is defined as (by other than medical reasons):
    * ≥ 45 years of age and has not had menses for >2 years
    * Amenorrheic for < 2 years without a hysterectomy and/or oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
    * Post hysterectomy or oophorectomy. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound.
14. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use two forms of highly effective contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) starting with the first dose of study therapy and to continue its use for 30 days after the last dose of study therapy, or abstain from heterosexual activity.

Exclusion Criteria:

1. Relapsed pure seminoma
2. Rising tumor markers (AFP and hCG) at time of screening
3. Patients who completed 2nd cycle of HDCT (time since last dose of HDCT) >16 weeks ago
4. Treatment with any investigational agent within 28 days prior to study registration
5. Other active malignancy requiring treatment in past 12 months
6. History of psychiatric illness or social situations that would limit compliance with study requirements
7. Active infection requiring systemic therapy
8. Previous hypersensitivity to etoposide which did not recover with supportive care
9. Pregnancy, lactation, or breastfeeding
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
12-month Progression Free Survival | time from the date of randomization to the date of disease relapse or death (i.e. up to 1 year)
  Investigator determination of tumor progression (clinical, radiographic, tumor markers including AFP and hCG)

SECONDARY OUTCOMES:
12-month Overall Survival | Time of registration to death from any cause (i.e. up to 1 year)
Assess toxicity and tolerability of maintenance etoposide | through study completion (i.e. up to 2 years)
  Toxicities according to CTCAE v5 will be summarized by frequencies and rates calculated as the proportion of patients in the safety population experiencing SAEs, discontinuations due to AEs, and AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Adra, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taza F, Abonour R, Zaid MA, Althouse SK, Anouti B, Akel R, Hanna NH, Adra N, Einhorn LH. Maintenance Oral Etoposide After High-Dose Chemotherapy (HDCT) for Patients With Relapsed Metastatic Germ-Cell Tumors (mGCT). Clin Genitourin Cancer. 2023 Apr;21(2):213-220. doi: 10.1016/j.clgc.2023.01.004. Epub 2023 Jan 18. PMID 36737276